CLINICAL TRIAL: NCT02386761
Title: A Phase 1, Randomised Double-blind, Placebo-controlled STUDY of Single and Repeated Ascending doseS in Healthy Volunteers to Investigate the Safety, Tolerability and Pharmacokinetics of Inhaled CHF 6001
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of Inhaled CHF6001
Acronym: CHF6001Ext
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-06001AA1-08
Record Dates: First submitted 2015-01-22; First posted 2015-03-12 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tanimilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Ascending Dose (SAD) (Experimental): * Dose 1 (SAD1): 6 inhalations of CHF 6001 400 µg giving a total dose of 2400 µg
  * Dose 2 (SAD2): 10 inhalations of CHF 6001 400 µg giving a total dose of 4000 µg
  * Dose 3 (SAD3): 12 inhalations of CHF 6001 400 µg giving a total dose of 4800 µg Placebo (P): the number of placebo inhalations will match that of the active CHF 6001 pertaining to the same dose period.
  In case the actual doses are modified, the number of inhalations will be adapted accordingly.
  Interventions: Drug: Single Ascending Dose (SAD)
- Multiple Ascending Dose (MAD) (Experimental): * Dose 1 (MAD1): Multiple doses of CHF 6001 - Total daily dose 2400 µg or placebo
  * Dose 2 (MAD2): Multiple doses of CHF 6001 - Total daily dose 4000 µg or placebo
  * Dose 3 (MAD3): Multiple doses of CHF 6001 - Total daily dose 4800 µg or placebo
  Duration 14 days b.i.d.
  Interventions: Drug: Multiple Ascending Dose (MAD)

INTERVENTIONS:
Drug: Single Ascending Dose (SAD)
  Other Names: CHF6001
  Arms: Single Ascending Dose (SAD)
Drug: Multiple Ascending Dose (MAD)
  Other Names: CHF6001
  Arms: Multiple Ascending Dose (MAD)

SUMMARY:
A phase I randomised, double-blind, placebo-controlled study of single and repeated ascending doses in healthy volunteers to investigate the safety, tolerability and pharmacokinetics of inhaled chf 6001.

DETAILED DESCRIPTION:
To assess the safety and tolerability of single and repeated ascending doses of CHF 6001 in healthy volunteers and to investigate the pharmacokinetic (PK) profile of CHF 6001 and its metabolites CHF 5956 and CHF 6095.

ELIGIBILITY:
Main Inclusion

* Subject's written informed consent obtained prior to any study-related procedure
* Male and female Caucasian healthy volunteers aged 18-55 years inclusive
* Vital signs:Subjects aged 18-45: Diastolic BP 40-90, Systolic BP 90-140 Subjects aged 45-55: Diastolic BP 40-90, Systolic BP 90-150 (as mean of three measures performed after at least 5 minutes of resting); checked at screening visit and Day -1
* 12-lead digitised Electrocardiogram (12-lead ECG) considered as normal (40≤Heart rate≤110bpm,120 ms ≤ PR ≤ 210 ms, QRS ≤ 120 ms, QTcF ≤ 450 ms for males and ≤ 470ms for females) checked at screening visit and Day -1
* Lung function measurements within normal limits: FEV1 > 80% of predicted normal value (according to the Global Lung Function Initiative, ERS Task Force Lung Function Reference Values (1,2) ) and FEV1/FVC ratio > 0.70

Main Exclusion:

* Pregnant or lactating women
* Clinically significant cardiac abnormalities
* Any clinically relevant abnormal laboratory values

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 0-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, MD, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Nottingham, UK, United Kingdom

REFERENCES:
- [Background] Jolling K, Abelo A, Luyckx N, Nandeuil MA, Govoni M, Cella M, Lindauer A. Concentration-QT Modeling Following Inhalation of the Novel Inhaled Phosphodiesterase-4 Inhibitor CHF6001 in Healthy Volunteers Shows an Absence of QT Prolongation. CPT Pharmacometrics Syst Pharmacol. 2019 Jul;8(7):460-468. doi: 10.1002/psp4.12405. Epub 2019 May 11. PMID 31077576
- [Result] Mariotti F, Govoni M, Lucci G, Santoro D, Nandeuil MA. Safety, tolerability, and pharmacokinetics of single and repeat ascending doses of CHF6001, a novel inhaled phosphodiesterase-4 inhibitor: two randomized trials in healthy volunteers. Int J Chron Obstruct Pulmon Dis. 2018 Oct 18;13:3399-3410. doi: 10.2147/COPD.S174156. eCollection 2018. PMID 30425469